CLINICAL TRIAL: NCT07175675
Title: Operative Treatment vs Treatment With Semi-occlusive Dressing - a Randomized, Controlled Trial on Finger Amputations
Brief Title: Operative Treatment vs Treatment With Semi-occlusive Dressing for Single Finger Amputations
Acronym: FINACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R25023
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Fingertips Traumatic Amputations; Finger Injuries; Finger; Finger Injury; Amputation, Traumatic; Amputation
Keywords: finger amputation; single finger amputation; single digit amputation
MeSH Terms: conditions — Finger Injuries; Amputation, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Tamai zone 1 operative (Active Comparator): operative treatment of surgeons choice
  Interventions: Procedure: Operative treatment of surgeons choice
- Tamai Zone 1 non-operative (Experimental): treatment with semi-occlusive film
  Interventions: Procedure: Semi-occlusive film
- Tamai zone 2 operative (Active Comparator): Operative treatment of surgeons choice
  Interventions: Procedure: Operative treatment of surgeons choice
- Tamai Zone 2 non-operative (Experimental): treatment with semi-occlusive film
  Interventions: Procedure: Semi-occlusive film
- Tamai Zone 3-4 operative (fingers II-V) (Active Comparator): Operative treatment of surgeons choice
  Interventions: Procedure: Operative treatment of surgeons choice
- Tamai Zone 3-4 non-operative (fingers II-V) (Experimental): treatment with semi-occlusive film
  Interventions: Procedure: Semi-occlusive film

INTERVENTIONS:
Procedure: Operative treatment of surgeons choice — treatment of single finger amputation with revision amputation, local or micro-vascular flap as best befits each specific injury
  Arms: Tamai Zone 3-4 operative (fingers II-V); Tamai zone 1 operative; Tamai zone 2 operative
Procedure: Semi-occlusive film — The film is placed on a cleansed wound surface. bone is shortened to the level of injury. Visible nerves, arteries and tendons are cut and allowed to retract. The film is to be changed once weekly until the wound has closed.
  Arms: Tamai Zone 1 non-operative; Tamai Zone 2 non-operative; Tamai Zone 3-4 non-operative (fingers II-V)

SUMMARY:
The goal of this interventional study is to find out whether conservative treatment with semi-occlusive film is superior to surgical treatment in single finger amputations in adult population. The main question it aims to answer is:

Is PRWHE (Patient Reported Wrist and Hand Evaluation) total score measured at 12 months after injury better in conservatively or operatively treated patients?

DETAILED DESCRIPTION:
The aim of this study is to compare the outcomes of operative treatment (chosen by the surgeon, including amputation revision with primary skin closure or flap coverage for the tissue defect) versus non-operative treatment using a semi-occlusive dressing for single finger amputations. This study is a randomized controlled superiority trial including three strata, each with two treatment arms, allocated in a 1:1 ratio. The three strata of the study design are based on the level of amputation as follows: Stratum 1 = Tamai Zone 1, Stratum 2 = Tamai Zone 2, Stratum 3 = Tamai Zones 3+4 (fingers II-V only). In all strata, the treatment arms are A (operative) and B (non-operative). Randomization will be performed as computer generated randomization with 1:1 allocation.

Primary objective is to determine whether treatment with semi-occlusive dressings is superior to operative treatment after a single finger amputation in each stratum, measured with PRWHE at 12 months after injury.

ELIGIBILITY:
Inclusion Criteria:

* age >18, single digit injury, Amputation at Tamai zones 1+2 in all digits or Tamai zones 3+4 in digits II-V, Able to understand Finnish and to complete self-reported questionnaires

Exclusion Criteria:

* Previous partial or total amputation of the injured digit, Previous condition which affects significantly the function and/or symptoms of the affected hand, Patient is pregnant at the time of recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
PRWHE | 12 months
  Our primary outcome measure is PRWHE mean difference (MD) between treatment arms in each stratum with the associated 95% confidence interval (CI) at 12 months post-randomization. Patient-Reported Wrist and Hand Evaluation (PRWHE) was chosen, because it covers both pain and loss of function which are the main symptoms after a digital amputation, has evidence of reliability, validity and responsiveness in hand and wrist trauma population, and is considered slightly more responsive than DASH. As a patient reported outcome, it is prone to ascertainment bias - especially since in this study setting it is not possible to blind the participant to given treatment. To overcome this, we have included several objective outcome measures as secondary outcomes. Nevertheless, Patient-Reported Outcome Measures are considered the most meaningful instruments for outcome evaluation in musculoskeletal conditions, because those assess patient-perceived important symptoms and disability.

SECONDARY OUTCOMES:
PRWHE 1 month | 1 month
  PRWHE mean difference (MD) between treatment arms in each stratum with the associated 95% confidence interval (CI) at 1 month post-randomization.
PRWHE 3 months | 3 months
  PRWHE mean difference (MD) between treatment arms in each stratum with the associated 95% confidence interval (CI) at 3 months post-randomization.
PRWHE 6 months | 6 months
  PRWHE mean difference (MD) between treatment arms in each stratum with the associated 95% confidence interval (CI) at 6 months post-randomization.
Return to daily activities 1 month | 1 month
  return to daily activities is collected at 1, 3, 6, and 12 months. Amputation injuries are significant indicators for being off work and having a prolonged time off work. Potential difference between treatment arms in Return to ordinary daily activities could have wider economic implications and work as a factor in determining the most beneficial treatment option for each patient.
Return to daily activities 3 months | 3 months
  return to daily activities is collected at 1, 3, 6, and 12 months. Amputation injuries are significant indicators for being off work and having a prolonged time off work. Potential difference between treatment arms in Return to ordinary daily activities could have wider economic implications and work as a factor in determining the most beneficial treatment option for each patient.
Return to daily activities 6 months | 6 months
  return to daily activities is collected at 1, 3, 6, and 12 months. Amputation injuries are significant indicators for being off work and having a prolonged time off work. Potential difference between treatment arms in Return to ordinary daily activities could have wider economic implications and work as a factor in determining the most beneficial treatment option for each patient.
Return to daily activities 12 months | 12 months
  return to daily activities is collected at 1, 3, 6, and 12 months. Amputation injuries are significant indicators for being off work and having a prolonged time off work. Potential difference between treatment arms in Return to ordinary daily activities could have wider economic implications and work as a factor in determining the most beneficial treatment option for each patient.
Michigan Hand Questionnaire (MHQ) aesthetics subsection 6 months | 6 months
  MHQ aesthetics subsection will be collected at 6 and 12 months. We will analyse a MD between treatment arms in each stratum with the associated 95% CI. Reliability, validity, and responsiveness of the MHQ is well-documented. Aesthetics is of interest to measure patient satisfaction with more than pain or function focused questionnaires.
Michigan Hand Questionnaire (MHQ) aesthetics subsection 12 months | 12 months
  MHQ aesthetics subsection will be collected at 6 and 12 months. We will analyse a MD between treatment arms in each stratum with the associated 95% CI. Reliability, validity, and responsiveness of the MHQ is well-documented. Aesthetics is of interest to measure patient satisfaction with more than pain or function focused questionnaires.
Cold Intolerance Symptom Severity (CISS) 6 months | 6 months
  We will analyse a MD between treatment arms in each stratum with the associated 95% CI. Cold intolerance is recognized as a disabling sequelae of upper extremity trauma, especially when neurovascular structures are involved. CISS test score ranges between a minimum of 4 and a maximum of 100, where lower is better.
Cold Intolerance Symptom Severity (CISS) 12 months | 12 months
  We will analyse a MD between treatment arms in each stratum with the associated 95% CI. Cold intolerance is recognized as a disabling sequelae of upper extremity trauma, especially when neurovascular structures are involved. CISS test score ranges between a minimum of 4 and a maximum of 100, where lower is better.
Patient Accepted Symptom State (PASS) 1 month | 1 month
  PASS is collected at 1, 3, 6 and 12 months. PASS will be assessed with the statement, "I am satisfied with the pain level and function of my finger/thumb," rated on a 5-point Likert scale (strongly disagree, somewhat disagree, neither agree nor disagree, somewhat agree, strongly agree). We will also assess whether the patients would choose the same treatment again with the statement "If I would be in the same circumstances, I would be willing to undergo this treatment again" rated on the same 5-point Likert scale as the previous statement. Results will be dichotomized between 'neither agree nor disagree' and 'somewhat agree' for both statements. This type of questionnaire has been shown to have good test-retest reliability and construct validity
Patient Accepted Symptom State (PASS) 3 months | 3 months
  PASS is collected at 1, 3, 6 and 12 months. PASS will be assessed with the statement, "I am satisfied with the pain level and function of my finger/thumb," rated on a 5-point Likert scale (strongly disagree, somewhat disagree, neither agree nor disagree, somewhat agree, strongly agree). We will also assess whether the patients would choose the same treatment again with the statement "If I would be in the same circumstances, I would be willing to undergo this treatment again" rated on the same 5-point Likert scale as the previous statement. Results will be dichotomized between 'neither agree nor disagree' and 'somewhat agree' for both statements. This type of questionnaire has been shown to have good test-retest reliability and construct validity
Patient Accepted Symptom State (PASS) 6 months | 6 months
  PASS is collected at 1, 3, 6 and 12 months. PASS will be assessed with the statement, "I am satisfied with the pain level and function of my finger/thumb," rated on a 5-point Likert scale (strongly disagree, somewhat disagree, neither agree nor disagree, somewhat agree, strongly agree). We will also assess whether the patients would choose the same treatment again with the statement "If I would be in the same circumstances, I would be willing to undergo this treatment again" rated on the same 5-point Likert scale as the previous statement. Results will be dichotomized between 'neither agree nor disagree' and 'somewhat agree' for both statements. This type of questionnaire has been shown to have good test-retest reliability and construct validity
Patient Accepted Symptom State (PASS) 12 months | 12 months
  PASS is collected at 1, 3, 6 and 12 months. PASS will be assessed with the statement, "I am satisfied with the pain level and function of my finger/thumb," rated on a 5-point Likert scale (strongly disagree, somewhat disagree, neither agree nor disagree, somewhat agree, strongly agree). We will also assess whether the patients would choose the same treatment again with the statement "If I would be in the same circumstances, I would be willing to undergo this treatment again" rated on the same 5-point Likert scale as the previous statement. Results will be dichotomized between 'neither agree nor disagree' and 'somewhat agree' for both statements. This type of questionnaire has been shown to have good test-retest reliability and construct validity
Standard two-point discrimination | 12 months
  Tests evaluating finger pulp sensitivity are frequently used in clinical practice. S2PD has been used in many digital nerve repair studies, and has good test retest and interobserver reliability, although has received criticism for lack of standardization in previous studies. S2PD normative results depend on the age of the patients, being close to 2mm in younger patients and around 4mm in elderly population. Generally, the lower the result, the better sensation is in the fingertip.
Moberg pick up test (MPUT) | 12 months
  MPUT is a standardized test designed to evaluate hand dexterity. Fine motor dexterity of the hand can be affected by disruptions in sensation of fingertips, meriting use of this outcome measure for this study. MPUT normative data depends on the age of the patient and is approximately 12 seconds for young patients (20-39yo) and 16-17 seconds for elderly patients (60+yo). Generally, the lower the result, the better.
Range of motion (ROM) | 12 months
  ROM is measured to reveal whether the remaining joints of the affected digit are regaining mobility or if there are limitations due to scar tissue, contractures, or stiffness. The functional range of motion is 19°-71° at the metacarpophalangeal, 23°-87° at proximal interphalangeal, and 10°-64° at distal interphalangeal joints.
Grip strength | 12 months
  Grip strength is measured using Jamar dynamometer, providing standardized, reliable data for comparisons. The closer the result is to that of the uninjured hand, the better.
Difference in bony length | 12 months
  X-rays are taken from the affected hand at baseline before any interventions and at 12-month follow-up to measure potential changes in bony length of the affected digit between treatment arms of each stratum

CONTACTS AND LOCATIONS:
Overall Officials: Jarkko Jokihaara, Professor, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere Univesity Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data is going to be analysed in pseudonymised form. Data can be shared outside the study group but within the EU and EEA area for this study's statistical analysis purpose only. The Data Safety Monitoring Committee has the right to review the data collected in the study and check that the study has been carried out in an appropriate manner. Individual participants cannot be recognized from the published results. The results are going to be published in peer-reviewed international medical journals. Summary statistics may be shared outside the study group if reasonable request is received - for example, for meta analysis purposes. No Identifying data will be shared outside the study group for any reason.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol will be published in an appropriate journal and it and ICF and SAP will be available from the publication date onward. Other IPD as described above will be available after the completion of the study.
Access Criteria: Summary statistics may be shared outside the study group if reasonable request is received - for example, for meta analysis purposes.